CLINICAL TRIAL: NCT06277570
Title: Investigation of the Effect of Superimposed Neuromuscular Electrical Stimulation With Active Contraction in Patients With Knee Osteoarthritis.
Brief Title: Investigation of the Effect of Superimposed Neuromuscular Electrical Stimulation in Patients With Knee Osteoarthritis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mustafa Ertuğrul Yaşa, Assistant Professor, Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-487
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Electric Stimulation Therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The sample of the study will consist of participants who applied to Etlik City Physical Therapy and Rehabilitation Hospital, were diagnosed with knee osteoarthritis by the physician, and will receive routine treatment in the electrotherapy unit. Patients will be randomly assigned to groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional physiotherapy (Active Comparator): Demographic and medical information of the patients (age, gender, height and body weight, occupation, educational status, CV, family history and surgical history, medical history related to knee osteoarthritis) and pain level will be questioned. Conventional physiotherapy modalities will be applied in the group; exercise training, hotpack, ultrasound and transcutaneous electrical nerve stimulation (TENS). Patients will be treated for one hour, three days a week, for eight weeks.
  The physical functions, muscle structure and knee joint cartilage thickness, quality of life and functional status of the patients will be evaluated before and after treatment.
  Interventions: Other: conventional physiotherapy
- NMES (Active Comparator): Demographic and medical information of the patients (age, gender, height and body weight, occupation, educational status, CV, family history and surgical history, medical history related to knee osteoarthritis) and pain level will be questioned. In addition to conventional physiotherapy methods, passive NMES treatment will be applied in the group.Patients will be treated for one hour, three days a week, for eight weeks.
  The physical functions, muscle structure and knee joint cartilage thickness, quality of life and functional status of the patients will be evaluated before and after treatment.
  Interventions: Other: conventional physiotherapy; Other: NMES
- superimposed NMES (Active Comparator): Demographic and medical information of the patients (age, gender, height and body weight, occupation, educational status, CV, family history and surgical history, medical history related to knee osteoarthritis) and pain level will be questioned. In addition to conventional physiotherapy methods, superimposed NMES treatment will be applied in the group. Patients will be treated for one hour, three days a week, for eight weeks.
  The physical functions, muscle structure and knee joint cartilage thickness, quality of life and functional status of the patients will be evaluated before and after treatment.
  Interventions: Other: conventional physiotherapy; Other: Superimposed NMES

INTERVENTIONS:
Other: conventional physiotherapy — Conventional physiotherapy is a treatment method that includes exercise training, hotpack, ultrasound and TENS (electrotherapy) applications.
Other: NMES — Neuromuscular Electrical Stimulation (NMES) is a non-invasive method that activates intramuscular nerve branches and produces visible contractions through surface electrodes placed on skeletal muscles.
  Arms: NMES
Other: Superimposed NMES — Superimposed NMES technique is the use of NMES with voluntary muscle contraction.
  Arms: superimposed NMES

SUMMARY:
The aim of the study is to investigate the effects of superimposed neuromuscular electrical stimulation with active contraction on physical function, muscle and joint structure, functionality, and quality of life in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a progressive joint disease that can affect all structures that make up the joint, especially cartilage. The frequency of OA increases with age and can especially affect weight-bearing joints such as the knee and hip joints. The main symptoms of knee OA are pain, decreased joint range of motion (ROM), decreased muscle strength, functional loss, and limitation in daily living activities. However, studies conducted in individuals with knee OA report a decrease in quadriceps muscle and knee joint cartilage thickness and impairment in sensorimotor function (proprioception and balance).

Many pharmacological and non-pharmacological methods are used in symptom management of knee OA. In this context, physiotherapy and rehabilitation are among the frequently used non-pharmacological methods. Exercise, manual therapy, taping, aqua therapy, thermal therapy, and electrotherapy are the basic physiotherapy modalities used in OA symptom management. Electrotherapy involves many different agents with different therapeutic purposes. One of these is Neuromuscular Electrical Stimulation (NMES). NMES is a non-invasive method that activates intramuscular nerve branches through surface electrodes placed on skeletal muscles and produces observable contractions. Although its most important therapeutic purpose is muscle stimulation, it also has contributions such as pain relief and sensory stimulation. Superimposed NMES technique (active NMES) is the use of NMES with voluntary muscle contraction. In superimposed NMES with active contraction, the patient is asked to actively contract the relevant muscle during each stimulation. Thus, exercise is performed simultaneously during electrotherapy application. When the literature is examined, there is no study investigating the effect of superimposed NMES with active contraction in patients with knee OA. In this context, the aim of this study is to investigate the effect of superimposed NMES with active contraction on physical function, muscle and joint structure, functionality and quality of life in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Having grade 2-3 knee osteoarthritis according to Kellgren and Lawrence Classification,
* Being between the ages of 40-65, ,
* Being literate
* Volunteer

Exclusion Criteria:

* Having Grade 2 or higher osteoarthritis in the hip, ankle, or foot joint Presence of a history of knee-related surgery (arthroplasty, meniscectomy, etc.)
* Having a deformity in the waist, leg, hip, knee, or ankle
* Having any inflammatory rheumatic, neurological, vestibular, cardiopulmonary disease
* Having active knee joint synovitis
* BMI>40
* Having a condition that is contraindicate for electrotherapy (malignancy, pacemaker, epilepsy, deep vein thrombosis, loss of protective sensation, etc.)
* Having received physiotherapy in the last 3 months
* Being diagnosed with a psychiatric disease
* Having a cooperation problem that makes it difficult to comply with evaluation and treatment

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | 8 weeks
  The muscle strength of the participants will be evaluated with a hand dynamometer. Before the measurements, participants will be placed in a sitting position on the bed with hips and knees flexed at 90º, feet free, arms crossed over the chest and without support. For the test, the participant will be asked to do maximum knee extension and at the last point, resistance will be given to disrupt the position with a hand dynamometer. When the test position is disrupted, the score seen on the dynamometer screen will be recorded.

SECONDARY OUTCOMES:
Joint position sense | 8 weeks
  The position sense of the knee joint will be evaluated with a digital inclinometer. Digital inclinometer is a motion-sensitive protractor. The test will be performed while the participants are in a prone position. Before the test, participants will be taught the target angle (20 degrees of flexion), and then they will be asked to reach this target angle again with their eyes closed. The amount of deviation from the target angle will be recorded as a score.
Muscle structure and knee joint cartilage thickness | 8 weeks
  Quadriceps muscle structure and knee joint cartilage structure will be evaluated with an ultrasonography device. Measurements will be taken from four sections of the quadriceps femoris muscle while the participants are at rest in the supine position. The measurement level will be determined as 50% of the femur length (the distance between the major trochanter and the lateral condyle). Muscle thicknesses will be determined by measuring the distance between the superficial and deep aponeurosis. The pennate angle will be calculated as the angle formed at the attachment point (insertion) of the muscle fascicles to the deep aponeurosis. Cartilage thickness will be measured at maximal knee flexion, in three regions: lateral, medial, and intercondylar.
Joint range of motion | 8 weeks
  Flexion and extension range of motion of the knee joint will be measured in degrees in the prone position using a goniometer. For measurement, the pivot point of the goniometer will be placed on the lateral condyle of the femur, its fixed arm will be placed on the lateral midline of the femur, and the movable arm of the goniometer will follow the fibula. The participant will be asked to actively bend and extend his knee and the final point value will be recorded as angle.
Short Form-36 | 8 weeks
  Participants' quality of life will be evaluated with Short Form-36. This scale is a 36-item survey that questions the individual's quality of life, considering the last 4 weeks. It has eight sections: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health, emotional wellbeing
Western Ontario and McMaster Universities Osteoarthritis Index Scale | 8 weeks
  The functional status of the participants will be measured using the Western Ontario and McMaster Universities Osteoarthritis Index Scale (WOMAC) scale. The scale, which consists of 24 questions, has 3 subsections: pain, stiffness and function. Higher scores indicate more severe symptoms, greater disability, and poorer health status.
Visual Analog Scale (VAS) | 8 weeks
  VAS is a horizontal line of 10 centimeters and the beginning of the line means no pain and the end of the line means unbearable pain. Participants will be asked to make a mark based on the pain they feel (9).
Balance assessment | 8 weeks
  Balance will be evaluated with the Balance Error Scoring System (BESS). This test is a short, easily administered static balance test. The test will be performed for 20 seconds in three different positions (double leg, single leg, tandem) on firm and foam surfaces. The number of balance deviations that occur in the participants during the test will be recorded as a score. High deviation score indicates more balance disorder.
Functional capacity | 8 weeks
  The 30-Second Chair Stand Test will be performed for functional capacity assessment. For this test, the participant will be seated in a chair without armrests and asked to sit and stand as much as possible for 30 seconds. The total number will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Ertuğrul YAŞA, Principal Investigator — Saglik Bilimleri Universitesi; Emre Adıgüzel, Study Director — Etlik City Hospital Physical Therapy and Rehabilitation Hospital; Oğuzhan METE, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Faculty of Physiotherapy and Rehabilitation, University of Health Sciences, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No